CLINICAL TRIAL: NCT06026683
Title: Conduction System Stimulation to Avoid Left Ventricle Dysfunction
Acronym: STAY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Ermengol Vallès, Principal investigator, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STAY trial
Record Dates: First submitted 2023-08-28; First posted 2023-09-07 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Atrioventricular Block, Second and Third Degree; Pacemaker-Induced Cardiomyopathy; Heart Failure
MeSH Terms: conditions — Atrioventricular Block; Neoplasm Metastasis; Heart Failure

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into 2 groups according to pacing site: CSP vs RVAP.
Who Masked: Participant, Outcomes Assessor
Masking Description: The study is blinded for the patient and for the echocardiographers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- CSP (Conduction system pacing) (Active Comparator): Patients with pacemaker implanted with conduction system pacing.
  Interventions: Device: Pacemaker implant
- RVAP (Right ventricular apical pacing) (Active Comparator): Patients with pacemaker implanted with right ventricular apical pacing.
  Interventions: Device: Pacemaker implant

INTERVENTIONS:
Device: Pacemaker implant — Implantation of pacemaker with conduction system pacing or right ventricular apical pacing

SUMMARY:
The aim of the study is to demonstrate that conduction system pacing (CSP) can preserve a normal ventricular function compared to right ventricular apical pacing (RVAP) in patients with pre-implant preserved left ventricular ejection fraction (LVEF) and a high burden of expected ventricular pacing due to atrioventricular conduction block (AV block).

After informed consent signature, patients with high degree AV block and normal LVEF will be randomized to permanent pacemaker stimulation with CSP vs RVAP.

All the patients have a complete evaluation before the procedure and at 3 and 6 months follow-up.

DETAILED DESCRIPTION:
The STAY trial (Conduction System sTimulation to Avoid left ventricle dYsfunction) is a single-center, prospective, randomized, parallel, controlled study, comparing mid-term outcomes in a population undergoing pacemaker implantation due to a high degree atrio-ventricular block (AVB). The study was approved by the Hospital Ethics Committee, in accordance with the Declaration of Helsinki. All patients signed informed consent and were implanted between September 2019 until December 2022 in a 1:1 randomized fashion to conventional RVAP vs CSP (HBS or LBBS). Randomization was performed during the pre-procedural antibiotic infusion.

All the patients have a complete evaluation before the procedure and at 3 and 6 months follow-up, including demographic and clinical characteristics, physical examination, twelve-lead ECG, Minnesota score (MLWHFQ), and blood test with NT-ProBNP determination. Patients also have a transthoracic echography before the procedure and at 6 months follow-up.

At 6 months echocardiographic and clinical data will be compared.

ELIGIBILITY:
Inclusion criteria:

1. Age of 18 years or more
2. Preserved or mild deteriorated LVEF (Simpson >40%) assessed by a recent (<1 month before implantation) transthoracic echocardiography.
3. Indication for pacing based on the presence of a high degree AVB, and consequently with an anticipated high burden of ventricular pacing (>50%).
4. Live expectancy of more than 6 months and capability to understand the protocol, signing the informed consent form and accomplish the follow-up.

Exclusion criteria:

1. Indication for implantable cardioverter defibrillator device.
2. Patients with previous LVD and a recovered LVEF
3. History of myocardial infarction/revascularization or cardiac surgery within 6 months before randomization
4. Pregnancy, active cancer treatment, or participation in another clinical trial with active treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Delta-LVEF at 6 months | 6 months
  Change in LVEF in each group at 6 months vs baseline LVEF

SECONDARY OUTCOMES:
Delta-LVEDD at 6 months | 6 months
  Change in Left ventricular end diastolic diameter (LVEDD) in each group at 6 months vs baseline LVEDD
Delta-MLWHFQ (Minnesota score) at 6 months | 6 months
  Change in MLWHFQ score in each group at 6 months vs baseline MLWHFQ score. The MLWHFQ score is obtained by using a questionnaire of 21 aspects. It depicts how heart failure affected the daily life of the patients during the last month previous to the questionnaire. Each question can be scored from 0 ("No" effect) to 5 ("Very much" effect)
Delta-New York Heart Association (NYHA) class at 6 months | 6 months
  Change in NYHA class in each group at 6 months vs baseline NYHA class. NYHA class places patients in one of four categories based on limitations of physical activity:
  * I: No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation or shortness of breath.
  * II: Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, shortness of breath or chest pain.
  * III: Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, shortness of breath or chest pain.
  * IV: Symptoms of heart failure at rest. Any physical activity causes further discomfort.
Delta-NTProBNP at 6 months | 6 months
  Change in NTProBNP levels in each group at 6 months vs baseline NTProBNP levels
Readmissions due to heart failure | 6 months
  Number of readmissions due to heart failure in each group during follow-up
New onset Atrial fibrillation | 6 months
  Number of new-onset atrial fibrillation episodes in each group during follow-up
Mortality | 6 months
  All-cause Mortality in each group during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Ermengol Vallès, PhD, Study Director — Parc de Salut Mar; Carlos González, M.D., Principal Investigator — Parc de Salut Mar. Universitat Autónoma de Barcelona.
Locations (1):
- Hospital del Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
Data will only be available upon reasonable request.

REFERENCES:
- [Derived] Gonzalez-Matos CE, Rodriguez-Queralto O, Zaraket F, Jimenez J, Casteigt B, Valles E. Conduction System Stimulation to Avoid Left Ventricle Dysfunction. Circ Arrhythm Electrophysiol. 2024 Feb;17(2):e012473. doi: 10.1161/CIRCEP.123.012473. Epub 2024 Jan 29. PMID 38284238